CLINICAL TRIAL: NCT04011956
Title: Prognosis and Integrative Assessment of Aortic Coarctation Patients in CHINA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Collaborators: Beijing Anzhen Hospital (Other); Bayi Children's Hospital Affiliated to PLA Army General Hospital, China (Other); Capital Institute of Pediatrics, China (Other)
Responsible Party: Sponsor
Other Study IDs: PICC
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Coarctation of Aorta
MeSH Terms: conditions — Aortic Coarctation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — If a blood specimen is obtained, it will be separated and stored at -80 ℃ as plasma, viable cells, and extracted DNA. If a saliva specimen is obtained, it is stored for DNA. If a tissue specimen is obtained, it will be cut into small pieces and stored at liquid nitrogen.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort of Aortic Coarctation: Patients diagnosed as aortic coarctation and undergone corrected procedures from 2002 to Feb 28th 2019 were recruited in Beijing Anzhen Hospital, recording the results of clinical lab and echocardiography.
- Perspective Cohort of Aortic Coarctation: Patients diagnosed as aortic coarctation and undergone corrected procedures after Mar. 1st 2019 will be recruited in Beijing Anzhen Hospital, recording the results of clinical lab and echocardiography.

SUMMARY:
This is a systemic research of Chinese aortic coarctation patients, aiming to determine risk factors and serial biomarkers of aortic coarctation in prognosis.

DETAILED DESCRIPTION:
The goal is to determine how much the left ventricle remodeling pre-operation and how it changes in the following-up duration after surgery, so does in the blood pressure and heart function. Risk factors associated with complications and prognosis are investigated and analyzed. Identification of novel biomarkers is needed to help predicting the prognosis, such as the left ventricle anti-remodeling, heart function and blood pressure improvement, as well as the exercise tolerance post-operation. The findings of this study will help the investigators developping new tests to monitor affected patients and optimize the operation as well as the follow-up procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of isolated coarctation of the aorta, or accompanied with atrial septal defect(ASD), ventricular septal defect (VSD), patent ductus arteriosus( PDA), patent foramen ovale (PFO);
* Patients who can cooperation with study procedures.

Exclusion Criteria:

* Co-morbidities that may independently affect cardiovascular function, including associated complicated congenital heart disease, such as hypoplastic left heart syndrome (HLHS), interruption of aortic arch (IAA), Shone Syndrome, moderate and severe mitral stenosis;
* History of known vasculopathy, genetic syndromes, diabetes mellitus, hyperlipoidemia or other cardiovascular risk factors.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with coarctation of the aorta, treated after 2002 in Beijing Anzhen Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular mass | Prior to primary treatment and during follow-up visit(one month to 20 years for retrospective cohort and one year for prospective cohort)
  Left ventricular mass will be measured by 2D echocardiography. For the retrospective cohort, the data is collected from the cases' medical record, and during follow-up visit.
Hypertension | one month to 20 years after primary treatment for retrospective cohort and one year after primary treatment for prospective cohort
  Both resting blood pressure and exercise-related blood pressure will be assessed for patients above 5 years old during the follow-up visit.

SECONDARY OUTCOMES:
Left ventricular systolic function | one month to 20 years after primary treatment for retrospective cohort and one year after primary treatment for prospective cohort
  Left ventricular systolic function assessed by echocardiography
Left ventricular diastolic function | one month to 20 years after primary treatment for retrospective cohort and one year after primary treatment for prospective cohort
  Left ventricular diastolic function assessed by echocardiography (TDI)
Left ventricular systolic heart function of longitudinal myocardium | one month to 20 years after primary treatment for retrospective cohort and one year after primary treatment for prospective cohort
  Left ventricular systolic heart function of longitudinal myocardium assessed by echocardiography (M mode Doppler).
Exercise tolerance | one month to 20 years after primary treatment for retrospective cohort and one year after primary treatment for prospective cohort
  Six minutes walking distance will be recorded and analyzed to evaluate the exercise tolerance. Echocardiographic images will be obtained after six minutes walking to assess the reserve function of left ventricle. Blood pressure will also be taken immediately after the Six minutes walking to analyze exercise-induced hypertension.
Biomarkers of vascular inflammation | Prior to primary treatment and during follow-up visit(one month to 20 years for retrospective cohort and one year for prospective cohort)
  Biomarkers of inflammation (hs-CRP). For the retrospective cohort, the data is collected from the cases' medical record, and during follow-up visit.
Biomarkers of left ventricle remodeling | For the retrospective cohort, follow-up visit of 1 month to 20 years after primary treatment. For the prospective cohort, the data is collected prior to primary treatment and during follow-up visit of one year after primary treatment
  Biomarkers of left ventricle remodeling (ST2)
Biomarkers of left heart function | Prior to primary treatment and during follow-up visit(one month to 20 years for retrospective cohort and one year for prospective cohort)
  Biomarkers of left heart function (BNP). For the retrospective cohort, the data is collected from the cases' medical record, and during follow-up visit.
Biomarkers of hypertension phenotype related to aortic coarctation | one month to 20 years after primary treatment for retrospective cohort and one year after primary treatment for prospective cohort
  Biomarkers of hypertension phenotype related to aortic coarctation
Recoarctation | one month to 20 years after primary treatment for retrospective cohort and one year after primary treatment for prospective cohort
  Recoarctation assessed by echocardiography or computed tomography angiography.
All-cause death | 20 years after primary treatment for retrospective cohort and one year after primary treatment for prospective cohort
  The data is collected during follow-up visit at follow-up time point.

CONTACTS AND LOCATIONS:
Overall Officials: Jie DU, PhD, Principal Investigator — Beijing Institute of Heart, Lung and Blood Vessel Diseases
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China